CLINICAL TRIAL: NCT01499212
Title: Effects of Different Inspiratory to Expiratory Ratios on Intrapulmonary Shunt Fraction and Oxygenation During One Lung Ventilation in the Lateral Decubitus Position
Brief Title: Effects of Different I:E Ratio on Intrapulmonary Shunt Fraction and Oxygenation During One Lung Ventilation in the Lateral Decubitus Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-2011-0058
Record Dates: First submitted 2011-12-18; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Lung Cancer; Lung Lobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I:E ratio 1:1 (Experimental)
  Interventions: Procedure: I:E ratio

INTERVENTIONS:
Procedure: I:E ratio — I:E ratio 1:1 Volume controlled ventilation TV:8ml/kg EtCO2:35-40mmHg

SUMMARY:
The purpose of this study is to investigate effect of increasing inspiratory time (I:E ratio 1:1) on intrapulmonary shunt fraction and oxygenation during one lung ventilation in the lateral decubitus position.

DETAILED DESCRIPTION:
Increasing inspiratory time(e.g. Inverse ratio ventilation) has been known that had advantage of alveolar recruitment, preventing of ateletasis. On the contrary, it has disadvantange of intrinsic PEEP, air trapping. There is few study on one lung ventilation in lateral decubitus position about this ventilation method. We were going to investigate effecf of this ventilation method.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I, II
* Use of Double lumen tube
* Unilateral lung lobectomy

Exclusion Criteria:

* COPD
* CAOD
* Unstable hemodynamic status
* Peak airway pressure > 30mmHg (Two lung ventilation)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
intrapulmonary shunt fraction | T1 (10min before one lung ventibation)T2 (30min after one lung ventilation started)T3 (60min after one lung ventilation started)T4 (10min after two lung ventilation)
  T1,T2,T3,T4 : ALL mesurement in lateral decubitus position T1-intrapulmonary shunt T2-intrapulmonary shunt T3-intrapulmonary shunt T4-intrapulmonary shunt

SECONDARY OUTCOMES:
Respiratory dynamic parameters | T1,T2,T3,T4 (same as primary outcome measure)
  Mechanical Ventilator measurement : Paw, Pplat, Pmean, Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, MD,PhD, Study Chair — Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Korea
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea